CLINICAL TRIAL: NCT06230198
Title: The Effect of Retrograde Autologous Priming on Transfusion Requirements After Cardiac Surgery (TheRAPy): a Multiple Period Vanguard Cluster Crossover Trial
Brief Title: The Effect of Retrograde Autologous Priming on Transfusion Requirements After Cardiac Surgery
Acronym: TheRAPy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: TheRAPy
Record Dates: First submitted 2023-12-23; First posted 2024-01-30 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Red Blood Cell Transfusion

STUDY DESIGN:
Intervention Model Description: a multiple period vanguard cluster crossover trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Retrograde autologous priming (Experimental): sites implement retrograde autologous priming (RAP) during cardiac surgery
  Interventions: Procedure: retrograde autologous priming (RAP)
- Crystalloid priming (Experimental): sites implement crystalloid priming use during cardiac surgery
  Interventions: Procedure: Crystalloid priming

INTERVENTIONS:
Procedure: retrograde autologous priming (RAP) — sites follow an institutional policy of routine use of retrograde autologous priming (RAP) during cardiac surgery
  Arms: Retrograde autologous priming
Procedure: Crystalloid priming — sites implement crystalloid priming use during cardiac surgery
  Arms: Crystalloid priming

SUMMARY:
The TheRAPy vanguard trial is a multicentre, multiple period randomized, cluster crossover vanguard trial testing the feasibility of a full-scale trial to evaluate whether a centre-based policy of routine use of RAP versus a policy of crystalloid priming reduces RBC transfusion for patients undergoing cardiac surgery on cardiopulmonary bypass. It will also provide information about key parameters of the TheRAPy full-scale trial.

DETAILED DESCRIPTION:
About 50% of patients undergoing cardiac surgery require red blood cell (RBC) transfusion. Given the limited blood supply and harms of transfusion, evidence-based blood conservation strategies are a priority. There is one such simple conservation technique called Retrograde autologous priming (RAP), in which the patient's own blood, rather than crystalloid fluid, is used to prime the heart-lung machine. Ultimately, it minimizes the loss of RBCs during surgery. Despite evidence of RAP reducing incidence of RBC transfusions by 40% and RBC units transfused by 38% in small randomized trials, it is not routinely used due to the uncertainty about overall benefit and potential harms. Routine RAP may be beneficial, but this needs to be confirmed in a large pragmatic randomized trial. Therefore, the goal of this vanguard trial is to assess the feasibility of a full-scale multi-centre randomized cluster crossover trial to determine whether an institutional policy of routine RAP reduces the number of RBC units transfused up to 72 hours after cardiac surgery compared to crystalloid priming. This will include 4 sites that will test the two policies in an alternating sequence during 12 periods of 4 weeks, with an expected volume of 4500 cardiac surgery patients. If the adherence to both polices is >=90%, a full trial will be conducted. The findings of this study have the potential to improve the outcomes of tens of thousands of patients around the world and will provide the basis for cardiac practice guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Hospitals completing >200 adult cardiac surgical cases a year; (ii) 95% of cardiovascular surgery group (i.e., cardiac anesthesiologists, surgeons, and perfusionists) agree to manage patients under both autologous priming policies as per their randomization schedule for the duration of the trial.
* All patients undergoing cardiac surgery on cardiopulmonary bypass at an enrolled site during the trial period will be included in data collection.

Exclusion Criteria:

* Complete <=200 cardiac surgical cases.
* <95% of their cardiovascular surgery group agrees to manage patients according to either of the two policies.

Ages: 10 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4500 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Feasibility of implementing a full-scale randomized cluster crossover trial | 6 months
  Feasibility is defined as adherence >90% to both institutional policies applied in random sequence.

SECONDARY OUTCOMES:
Data Collection about Critical Parameters | 6 months
  to collect data about critical parameters that affect the design and implementation of the full-scale trial

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Spence, MD, PhD, Principal Investigator — Population Health Research Institute
Locations (4):
- Canada (4):
  - St. Boniface Hospital, Winnipeg, Manitoba
  - Hamilton General Hospital, Hamilton, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No